CLINICAL TRIAL: NCT06522789
Title: Could Automated Objective Measurements Acquired at the Preoperative Stage Estimate the Corrected Distance Visual Acuity After Corneal Cross-linking in Keratoconus?
Brief Title: Preoperative Corneal Measurements Estimate the Corrected Distance Visual Acuity After Corneal Cross-linking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sistina Ophthalmology Hospital (Other)
Responsible Party: Principal Investigator, Fanka Gilevska, Principal investigator, Sistina Ophthalmology Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 17-25 10.02.2017
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Keratoconus
Keywords: Keratoconus; cross-linking; corneal optical density
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator): The total number of patients who underwent CXL was seventy-seven; 23 were females, and 54 were males of the mean (±sd, range) age 24.2 (±7.0, 11-44) years.
  Interventions: Procedure: corneal cross-linking procedure
- Group 2 (No Intervention): Twenty-three patients, six females and 17 males of mean age 27.3 (±7.0, 17-44) years, were untreated.
- Group 3 (No Intervention): Twenty-four subjects, nine females and 15 males of mean age 24.7 (±7.6, 17-45) years, were recruited as controls.

INTERVENTIONS:
Procedure: corneal cross-linking procedure — Standard Dresden protocol corneal cross-linking procedure The CXL procedure adhered to the standard Dresden protocol. All patients received topical anaesthetic (Tetracaine HCL 0.5%, Alcon Forth Worth, Texas) and a miotic (Isopto Carpine 2% HCl, Alcon, Fort Worth, Texas) drops 30 minutes before the procedure. The periocular region and conjunctival sac were washed with 10% povidone-iodine (Betadine 10%, Alcaloid, Skopje). Manual epithelial scraping with a crescent knife followed. Pachymetry was kept over 400 μm during the procedure and measured with an ultrasound hand pachymeter (Pocket II, Quantel Medical, Cournon d'Auvergne, France). Riboflavin (Peschke D, Peschke Trade, Huenenberg, Switzerland) was applied every 3 minutes for 30 minutes. We performed corneal UV-A radiation with a wavelength of 370 nm and energy of 3mW using a UVA CXL lamp (VEGA CBM-X-Linker, Carleton Optical, Chesham, UK) for 30 minutes (6 cycles of 5 minutes each).
  Arms: Group 1

SUMMARY:
This study aims to determine if objective markers describing corneal optical density (COD), thinnest corneal thickness (TCT), anterior (ARC), and posterior (PRC) surface radii over the 3mm thinnest region of the cornea could provide a model for calculating corrected distance visual acuity (CDVA) after corneal cross-linking (CXL) in keratoconus.

DETAILED DESCRIPTION:
A prospective, partially masked, semi-randomised, interventional clinical trial was undertaken between April 2018 and July 2023 in the refractive surgery department of the Sistina Ophthalmology Hospital in Skopje.

The patients' examination before the treatment and on every follow-up was a meticulous process that included assessment of CDVA (Aitomu LCD Digital Vision Eye Chart, Shanghai, China), refraction, tonometry, and corneal characteristics using Pentacam HR (Oculus, Optikgeräte GmbH, Wetzlar, Germany), biomicroscopy and dilated fundus examination. Corneal topography, thickness distribution, and COD profiles were captured for later analysis. The COD profile, which describes the turbidity of the cornea in the central apical region and the three concentric annular zones, was a vital part of the examination. The Pentacam software computed a figure, ranging from 0 (totally clear) to 100 (totally opaque), along a grey scale describing the optical density in each of the 12 regions. A higher number signifies increased turbidity and reduced transparency; a lower number represents the opposite. The software also averaged the total optical density in the apex, each concentric zone, each layer, and the cornea. A total of 20 COD values are generated for a single cornea. COD values for the central 0-2mm region covering the anterior (0-2ant) and central layers (0-2cent), paracentral 2-6mm annulus covering the anterior (2-6ant) and central layers (2-6cent), total anterior region layer (tot ant), total central layer (tot cent), and whole cornea (tot) were recorded. Separate COD values for the peripheral (6-10mm and 10-12mm annuli) and posterior (60µ) regions of the cornea were excluded as these regions are least likely to be affected by CXL. On all occasions, three consecutive Pentacam scans were taken in a dark room, and the best-quality scan was selected for recording and analysis. For each case, the COD (in greyscale units), thinnest corneal thickness (TCT, µ), anterior (ARC) and posterior (PRC) corneal radii of curvature(mm) values measured over a 3mm diameter zone covering the cone of the cornea were sequestered from the best scan.

The CXL procedure for group one adhered to the standard Dresden protocol. All patients received topical anaesthetic (Tetracaine HCL 0.5%, Alcon Forth Worth, Texas) and a miotic (Isopto Carpine 2% HCl, Alcon, Fort Worth, Texas) drops 30 minutes before the procedure. The periocular region and conjunctival sac were washed with 10% povidone-iodine (Betadine 10%, Alcaloid, Skopje). Manual epithelial scraping with a crescent knife followed. Pachymetry was kept over 400 μm during the procedure and measured with an ultrasound hand pachymeter (Pocket II, Quantel Medical, Cournon d'Auvergne, France). Riboflavin (Peschke D, Peschke Trade, Huenenberg, Switzerland) was applied every 3 minutes for 30 minutes. We performed corneal UV-A radiation with a wavelength of 370 nm and energy of 3mW using a UVA CXL lamp (VEGA CBM-X-Linker, Carleton Optical, Chesham, UK) for 30 minutes (6 cycles of 5 minutes each). Device testing was performed before every procedure, and irradiance density measured between 2.7-and-3.3 mW/cm2 was tolerated. At the end of the corneal CXL procedure, topical atropine 1% (Atropine Sulphate, Cooper, Athens, Greece), antibiotic (Tobrex, Alcon, Fort Worth, Texas) drops were instilled and a bandage soft contact lens (Air Optix Night & Day Aqua, Alcon, Texas) was placed over the cornea. Peschke® D. Riboflavin used in the study group was a standard Riboflavin solution consisting of 0.1% Riboflavin diluted into 20% dextran 500. The soaking time was 20-30 minutes or until microscopy showed riboflavin particles in the anterior chamber. Tobradex (Alcon, Fort Worth, Texas) eyedrops, a suspension of 0.3% Tobramycine and 0.05% Dexamethasone were prescribed for application after CXL. The dosage was four times per day for the first two weeks, then tapered twice daily for the next two weeks, and then to one drop per day for the last two weeks. All patients received topical steroids for a total of 6 weeks.

The postoperative care was comprehensive, ensuring the patient's well-being and recovery. It included a combination of antibiotic/corticosteroid drops instilled four times daily for the next two weeks, after which the drops were tapered off gradually over six weeks. Postoperative examinations were scheduled for one day, four days, 1-week until epithelisation and bandage lens removal, then 1-,3-,6-months, and 1-year postoperatively. After that, the patients were advised to complete an ophthalmological examination at least yearly.

Data from the treated eye, or just the right eye in bilateral cases, were analysed. Details of CDVA, COD, TCT, ARC and PRC values were stored in Excel (Microsoft, Redmond, WA) and analysed to determine the significance of any differences between groups (Mann Whitney U test or unpaired t-test) and changes occurring within each group (Friedman test or 1-way ANOVA for repeat measures, Wilcoxon signed rank or paired t-test). If significant changes were found, then the analysis would be extended to determine the significance of any association between the change (i.e., preop value-postop value) in the parameter and the value at the start of the study (Spearman's rho or Pearson correlation). Depending on the outcome of this analysis, the data would be further scrutinised to determine if a feasible model could be constructed (linear and multiple regression analysis) to predict the likely CDVA after CXL or after one year in untreated cases. Non-parametric tests were applied when data were not normally distributed (Kolmogorov-Smirnov test of normality). The changes and differences were considered statistically significant when p˂0.05.

ELIGIBILITY:
Inclusion Criteria:

Group 1 consisted of cases in which the astigmatism had increased by 1D or more, according to subjective refraction and corneal surface topography, over the previous year.

* Group 2 subjects consisted of confirmed keratoconus without signs of progression who opted to continue with their prescription glasses and tear-enhancing drops where necessary
* Group 3 is a control group of age- and gender-matched individuals without signs of keratoconus.

Exclusion Criteria:

* prior corneal surgeries, pachymetry less than 400 microns, scars or cloudings of the cornea, chemical injuries, severe dry eye, delayed epithelial healing and any inflammatory eye surface process before the CXL procedure

Ages: 11 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 124 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Association between preoperative corneal characteristics derived by Pentacam and subjective parameter CDVA and postoperative CDVA at the end of the follow-up period | one year
  Associations between Corneal Optical Density, Thinnest Corneal Thickness, Anterior Radius Curvature (ARC), Posterior Radius Curvature (PRC), ARC/PRC ratio, CDVA values at the start of the study and CDVA at postoperative.
Associations between predicted and actual CDVA following CXL | one year
  The differences in the mean predicted values measured at six months and one year.

SECONDARY OUTCOMES:
Corrected Distance Visual Acuity (CDVA) changes in all three groups during the follow up | one year
  Comparison of CDVA changes between the groups
Corneal Optical Density (COD) changes in all three groups during the follow up | one year
  COD values for the central 0-2mm region covering the anterior (0-2ant) and central layers (0-2cent), paracentral 2-6mm annulus covering the anterior (2-6ant) and central layers (2-6cent), total anterior region layer (tot ant), total central layer (tot cent), and whole cornea (tot) were recorded. Separate COD values for the peripheral (6-10mm and 10-12mm annuli) and posterior (60µ) regions of the cornea were excluded as these regions were least likely to be affected by CXL.
Corneal thickness (TCT) changes in all three groups during the follow up. | one year
  Comparison of TCT changes between the groups

CONTACTS AND LOCATIONS:
Overall Officials: Fanka Gilevska, PhD cand, Principal Investigator — Sistina Ophthalmology Hospital
Locations (1):
- Fanka Gilevska, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilevska F, Biscevic A, Bohac M, Patel S. Could Automated Objective Measurements Acquired at the Preoperative Stage Estimate the Corrected Distance Visual Acuity after Corneal Cross-Linking in Keratoconus? Ophthalmol Ther. 2024 Oct;13(10):2599-2614. doi: 10.1007/s40123-024-00993-0. Epub 2024 Aug 7. PMID 39110318